CLINICAL TRIAL: NCT05692895
Title: Immunohistochemical Expression of PDL1 In Primary Colorectal Carcinoma and Its Prognostic Impact
Brief Title: PDL1 In Primary Colorectal Carcinoma and Its Prognostic Impact
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Amira Ahmed Abdelnaby, Lecturer of pathology, Sohag University
Other Study IDs: Soh-Med-22-12-36
Record Dates: First submitted 2023-01-11; First posted 2023-01-20 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: PDL1- Colorectal Carcinoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Colorectal cancer (CRC) is a highly heterogenous disease. It the third most commonly diagnosed cancer in the world and the second cause of death among cancer cases mortality. Its incidence is rising all over the world, especially in developing countries . In Egypt it is coming the seventh cancer in incidence according to World Health Organization (WHO, 2020). Although there is much improvement in the diagnosis and treatment, but CRC is still constituting a big impact on human life and health, so researchers are trying to find out new therapeutic targets .

Programmed cell death protein 1 (PD-1) is an inhibitory receptor which is expressed on the surface of T lymphocytes during activation. Its role is to control T cell effector activity for various cellular responses as infections, autoimmune reactions, and cancer .

Cancer cells develop PD-ligand1 (PD-L1) expression which is a transmembrane molecule belonging to B7 family. Its action is through PD-1/PD-L1 reaction, and causing invasion and metastasis of cancer cells by protecting it from immunosurveillance by inhibiting T cell effector function, leading to carcinogenesis and development of many cancers including colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Both endoscopic and excisional biopsy specimens.
2. All the studied cases include sufficient materials for the immunohistochemical study.
3. Complete clinical data

Exclusion Criteria:

1. Patients with recurrence of the primary tumor.
2. Patients with a history of preoperative chemotherapy and/or radiotherapy.
3. Insufficient or tiny tissue biopsies

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A retrospective study will be carried out on 60 colorectal carcinoma specimens that were collected randomly from archives of Pathology Department, Faculty of Medicine, Sohag University
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-02 (Estimated); Primary Completion 2023-04 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Diagnosis and prognosis of colorectal carcinoma | Two or three days after staining tissue sections with PDL1 antibody
  Immunohistochemical expression of PDL1 in primary colorectal carcinoma

CONTACTS AND LOCATIONS:
Overall Officials: Amira A Abdelnaby, Lecturer, Principal Investigator — Faculty of medicine ,Sohag university

IPD SHARING:
Plan to Share IPD: Undecided